CLINICAL TRIAL: NCT02100878
Title: Effect of Exercise on the Neural Response to Food Cues and Energy Intake in Lean and Obese Adolescents
Brief Title: Exercise and Neural Response to Food Cues in Children
Status: Withdrawn | Type: Observational
Sponsor: Université Blaise Pascal, Clermont-Ferrand (Other)
Responsible Party: Principal Investigator, THIVEL David, Research Scientist, Université Blaise Pascal, Clermont-Ferrand
Other Study IDs: AU1107
Record Dates: First submitted 2014-03-27; First posted 2014-04-01 (Estimated); Last update posted 2014-04-02 (Estimated); Status verified 2014-04

CONDITIONS: Exercise Condition (EX); Control Session (CON)

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Lean adolescents
- Obese adolescents

SUMMARY:
Physical exercise has been shown to significantly reduce subsequent energy intake in obese adolescents but not in lean, without altering their appetite feelings. Although previous studies have pointed out the role of gastric peptides in this post exercise nutritional response, some recent work question the role of the neural system in the post exercise drive to eat. This study tends to explore whether or not an acute bout of exercise can affect the neural response to food cues in adolescents, obese or lean.

DETAILED DESCRIPTION:
After a medical inclusion, the adolescents will have to realise a DXA to assess their body composition and a submaximal exercise to evaluate their aerobic capacities.

They will have then to enter the laboratory on 2 different occasions in a randomized order from 8am to 330pm: At 8am they will receive a calibrated breakfast. then, at 1045; they will have to complete one of the experimental condition: 1) a cycling exercise or 2) remaining sitting fpr one hour. after the one hour sitting station or the exercise bout, they will be asked to complete a computer task while and electroencephalogram will be recorded. This computer task consists in visual recognition of rare pictures compared to frequent ones (oddball method). at 1215 they will be offered ad libitum meals. At regular intervals through the day, their appetite feelings will be assessed using Visual analogue scales.

Ad libitum energy consumption will be assessed by investigators and recorded for each participants.

ELIGIBILITY:
Inclusion Criteria:

* male
* 12-15 years old
* BMI defining obesity (Cole et al., 2000)
* Not being under diet restriction
* Information and consent forms have to be signed by the adolescent and his legal representative
* being registered to the national social security system

Exclusion Criteria:

* Being under medication
* contraindication to exercise
* smokers
* dieting

Ages: 12 Years to 15 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Lean and obese adolescents will be recruited accodring to the international curves for obesity. they will be between 12 to 15 years old and will have no medical limitations to complete exercise testings.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2014-03; Primary Completion 2014-03 (Actual); Study Completion 2015-03 (Estimated)

PRIMARY OUTCOMES:
Neural response to food cues | up to 2 months
  The electroencephalogram signals amplitude in response to visual food cues will be the primary outcome, after the exercise (during the exercise condition) and after the sitting position (during the control session)

CONTACTS AND LOCATIONS:
Locations (1):
- Laboratory AME2P, Aubière, France